CLINICAL TRIAL: NCT03387085
Title: NANT Triple Negative Breast Cancer (TNBC) Vaccine: Molecularly Informed Integrated Immunotherapy Combining Innate High-affinity Natural Killer (haNK) Cell Therapy With Adenoviral and Yeast-based Vaccines to Induce T-cell Responses in Subjects With TNBC Who Have Progressed on or After Standard-of-care Therapy.
Brief Title: QUILT-3.067: NANT Triple Negative Breast Cancer (TNBC) Vaccine: Molecularly Informed Integrated Immunotherapy in Subjects With TNBC Who Have Progressed on or After Standard-of-care Therapy.
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study halted prematurely and will not resume; participants are no longer being examined or receiving intervention
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.067
Record Dates: First submitted 2017-12-21; First posted 2017-12-29 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Triple Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — ALT-803; yeast-CEA vaccine; avelumab; Bevacizumab; Capecitabine; Cisplatin; Cyclophosphamide; Fluorouracil; Leucovorin; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NANT triple negative breast cancer (TNBC) Vaccine (Experimental): A combination of agents will be administered to subjects in this study: Aldoxorubicin HCl, N-803, ETBX-011, ETBX-051, ETBX-061, GI-4000, GI-6207, GI-6301, haNK, avelumab, bevacizumab, capecitabine, cisplatin, cyclophosphamide, 5-fluorouracil, leucovorin, nab-paclitaxel, SBRT.
  Interventions: Drug: Aldoxorubicin HCl; Biological: N-803; Biological: ETBX-011; Biological: ETBX-051; Biological: ETBX-061; Biological: GI-4000; Biological: GI-6207; Biological: GI-6301; Biological: haNK for Infusion; Biological: avelumab; Biological: bevacizumab; Drug: Capecitabine; Drug: Cisplatin; Drug: Cyclophosphamide; Drug: 5-Fluorouracil; Drug: Leucovorin; Drug: nab-Paclitaxel; Procedure: SBRT

INTERVENTIONS:
Drug: Aldoxorubicin HCl — Aldoxorubicin hydrochloride
Biological: N-803 — Recombinant human super agonist interleukin-15 (IL-15) complex
Biological: ETBX-011 — Ad5 [E1-, E2b-]-CEA
Biological: ETBX-051 — Ad5 [E1-, E2b-]-Brachyury vaccine
Biological: ETBX-061 — Ad5 [E1-, E2b-]-MUC1
Biological: GI-4000 — Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Ras proteins
Biological: GI-6207 — Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant CEA proteins
Biological: GI-6301 — Vaccine derived from recombinant Saccharomyces cerevisiae yeast expressing mutant Brachyury yeast proteins
Biological: haNK for Infusion — NK-92 [CD16.158V, ER IL-2]
Biological: avelumab — Recombinant human anti-PD-L1 IgG1 monoclonal antibody
Biological: bevacizumab — Recombinant human anti-VEGF IgG1 monoclonal
Drug: Capecitabine — 5'-deoxy-5-fluoro-N-[(pentyloxy) carbonyl]-cytidine
Drug: Cisplatin — cis-diamminedichloroplatinum(II)
Drug: Cyclophosphamide — 2-[bis(2-chloroethyl)amino]tetrahydro-2H-1,3,2-oxazaphosphorine 2-oxide monohydrate
Drug: 5-Fluorouracil — 5-fluoro-2,4 (1H,3H)-pyrimidinedione
Drug: Leucovorin — L-Glutamic acid, N-[4-[[(2-amino-5-formyl-1,4,5,6,7,8-hexahydro-4-oxo-6-pteridinyl)methyl]amino]benzoyl]-, calcium salt
Drug: nab-Paclitaxel — Benzenepropanoic acid, β-(benzoylamino)-α-hydroxy-(2aR, 4S, 4aS, 6R, 9S, 11S, 12S, 12aR, 12bS)-6,12b-bis(acetyloxy)-12-(benzoyloxy)-2a, 3, 4, 4a, 5, 6, 9, 10, 11, 12, 12a, 12b-dodecahydro-4,11-dihydroxy-4a, 8, 13, 13-tetramethyl-5-oxo-7,11-methano-1H-cyclodeca[3,4]benz[1,2-b]oxet-9-y1ester,(αR,βS)-(9CI) bound to albumin
Procedure: SBRT — Stereotactic Body Radiation Therapy

SUMMARY:
This is a phase 1b/2 study to evaluate the safety and efficacy of metronomic combination therapy in subjects with TNBC who have progressed on or after previous SoC chemotherapy. Phase 2 will be based on Simon's two-stage optimal design.

DETAILED DESCRIPTION:
Treatment will be administered in two phases, an induction and a maintenance phase, as described below. Subjects will continue induction treatment for up to 1 year. Treatment in the study will be discontinued if the subject experiences progressive disease (PD) or unacceptable toxicity (not corrected with dose reduction), withdraws consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment. Those who have a complete response (CR) in the induction phase will enter the maintenance phase of the study. Subjects who experience ongoing stable disease (SD) or an ongoing partial response (PR) at 1 year may enter the maintenance phase at the Investigator's discretion. Subjects may remain on the maintenance phase of the study for up to 1 year. Treatment will continue in the maintenance phase until the subject experiences PD or unacceptable toxicity (not corrected with dose reduction), withdraws consent, or if the Investigator feels it is no longer in the subject's best interest to continue treatment. The maximum time on study treatment, including both the induction and maintenance phases, is 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Able to understand and provide a signed informed consent that fulfills the relevant IRB or Independent Ethics Committee (IEC) guidelines.
3. Histologically-confirmed metastatic or unresectable TNBC that has either progressed on or after anthracycline-based chemotherapy (or other approved standard of care therapy) or subject has refused anthracycline-based chemotherapy, or other taxane- and platinum-based therapies. TNBC is defined as breast cancer that lacks estrogen receptor (ER) and progesterone receptor (PR) expression, and human epidermal growth factor receptor 2 (HER2) overexpression and/or amplification.
4. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2.
5. Have at least 1 measurable lesion of ≥ 1.0 cm.
6. Must have a recent formalin-fixed, paraffin-embedded (FFPE) tumor biopsy specimen following the conclusion of the most recent anticancer treatment. If an historic specimen is not available, the subject must be willing to undergo a biopsy during the screening period, if considered safe by the Investigator. If safety concerns preclude collection of a biopsy during the screening period, a tumor biopsy specimen collected prior to the conclusion of the most recent anticancer treatment may be used.
7. Must be willing to provide blood samples prior to the start of treatment on this study.
8. Must be willing to provide a tumor biopsy specimen 8 weeks after the start of treatment, if considered safe by the Investigator.
9. Ability to attend required study visits and return for adequate follow-up, as required by this protocol.
10. Agreement to practice effective contraception for female subjects of child-bearing potential and non-sterile males. Female subjects of child-bearing potential must agree to use effective contraception for up to 1 year after completion of therapy, and non-sterile male subjects must agree to use a condom for up to 4 months after treatment. Effective contraception includes surgical sterilization (eg, vasectomy, tubal ligation), two forms of barrier methods (eg, condom, diaphragm) used with spermicide, intrauterine devices (IUDs), and abstinence.

Exclusion Criteria:

1. Serious uncontrolled concomitant disease that would contraindicate the use of the investigational drug used in this study or that would put the subject at high risk for treatment-related complications.
2. Systemic autoimmune disease (eg, lupus erythematosus, rheumatoid arthritis, Addison's disease, autoimmune disease associated with lymphoma).
3. History of organ transplant requiring immunosuppression.
4. History of or active inflammatory bowel disease (eg, Crohn's disease, ulcerative colitis).
5. Inadequate organ function, evidenced by the following laboratory results:

   1. Absolute neutrophil count < 1000 cells/mm3.
   2. Platelet count < 75,000 cells/mm3.
   3. Uncorrectable grade 3 anemia (hemoglobin < 8 g/dL).
   4. Total bilirubin greater than the upper limit of normal (ULN; unless the subject has documented Gilbert's syndrome).
   5. Aspartate aminotransferase (AST [SGOT]) or alanine aminotransferase (ALT [SGPT]) > 2.5 × ULN (> 5 × ULN in subjects with liver metastases).
   6. Alkaline phosphatase levels > 2.5 × ULN (> 5 × ULN in subjects with liver metastases, or >10 × ULN in subjects with bone metastases).
   7. Serum creatinine > 2.0 mg/dL or 177 μmol/L.
   8. Serum anion gap > 16 mEq/L or arterial blood with pH < 7.3.
6. Uncontrolled hypertension (systolic > 160 mm Hg and/or diastolic > 110 mm Hg) or clinically significant (ie, active) cardiovascular disease, cerebrovascular accident/stroke, or myocardial infarction within 6 months prior to first study medication; unstable angina; congestive heart failure of New York Heart Association grade 2 or higher; or serious cardiac arrhythmia requiring medication. Subjects with uncontrolled hypertension should be medically managed on a stable regimen to control hypertension prior to study entry.
7. Serious myocardial dysfunction defined by ECHO as absolute left ventricular ejection fraction (LVEF) 10% below the institution's lower limit of predicted normal.
8. Dyspnea at rest due to complications of advanced malignancy or other disease requiring continuous oxygen therapy.
9. Positive results of screening test for human immunodeficiency virus (HIV).
10. Current chronic daily treatment (continuous for > 3 months) with systemic corticosteroids (dose equivalent to or greater than 10 mg/day methylprednisolone), excluding inhaled steroids. Short-term steroid use to prevent IV contrast allergic reaction or anaphylaxis in subjects who have known contrast allergies is allowed.
11. Known hypersensitivity to any component of the study medication(s).
12. Subjects taking any medication(s) (herbal or prescribed) known to have an adverse drug reaction with any of the study medications.
13. Concurrent or prior use of a strong cytochrome P450 (CYP)3A4 inhibitor (including ketoconazole, itraconazole, posaconazole, clarithromycin, indinavir, nefazodone, nelfinavir, ritonavir, saquinavir, telithromycin, voriconazole, and grapefruit products) or strong CYP3A4 inducers (including phenytoin, carbamazepine, rifampin, rifabutin, rifapentin, phenobarbital, and St John's Wort) within 14 days before study day 1.
14. Concurrent or prior use of a strong CYP2C8 inhibitor (gemfibrozil) or moderate CYP2C8 inducer (rifampin) within 14 days before study day 1.
15. Participation in an investigational drug study or history of receiving any investigational treatment within 30 days prior to initiation of treatment on this study, except for testosterone-lowering therapy in men with prostate cancer.
16. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol.
17. Concurrent participation in any interventional clinical trial.
18. Pregnant and nursing women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2024-01-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chan Soon-Shiong Institute for Medicine, El Segundo, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only the Phase 1b portion of the study enrolled participants. The study was terminated early, so no participants were enrolled on the Phase 2 portion of the study.
  Eligible participants could have gone through both induction and maintenance treatment on study.
Groups:
- NANT Triple Negative Breast Cancer (TNBC) Vaccine: A combination of agents was planned to be administered to subjects in this study: Aldoxorubicin HCl, N-803, ETBX-011, ETBX-051, ETBX-061, GI-4000, GI-6207, GI-6301, haNK, avelumab, bevacizumab, capecitabine, cisplatin, cyclophosphamide, 5-fluorouracil, leucovorin, nab-paclitaxel, SBRT.
Period: Overall Study
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
Started | 9
Completed | 2
Not Completed | 7
Not completed — Reason for Treatment Discontinuation | 7

BASELINE CHARACTERISTICS:
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.0 (6.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 2
subjects with TNBC who have progressed on or after previous SoC chemother [Count of Participants; unit: Participants] | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (AEs) and Serious AEs (SAEs)
Description: Graded using the NCI CTCAE Version 4.03.
Time Frame: Up to 2 years
Measure: Count of Participants; unit: Participants
Groups:
- NANT Triple Negative Breast Cancer (TNBC) Vaccine: A combination of agents were administered to subjects in this study: Aldoxorubicin HCl, N-803, ETBX-011, ETBX-051, ETBX-061, GI-4000, GI-6207, GI-6301, haNK, avelumab, bevacizumab, capecitabine, cisplatin, cyclophosphamide, 5-fluorouracil, leucovorin, nab-paclitaxel, SBRT.
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
Number analyzed (Participants) | 9
Participants
  Treatment emergent adverse events | 9
  Treatment emergent Serious Adverse Events | 5

2. Secondary Outcome: Objective Response Rate by RECIST v1.1
Description: Tumors will be assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase by computed tomography (CT) or magnetic resonance imaging (MRI) of target and non-target lesions in accordance with Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1. Percent of subjects with confirmed complete Response (CR; disappearance of all target lesions) or partial response (PR; >=30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum diameters.
Time Frame: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until confirmed disease progression. Up to 2.5 years
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
Number analyzed (Participants) | 9
Participants | 5

3. Secondary Outcome: Objective Response Rate by irRC (Percent of Subjects With Confirmed Complete or Partial Overall Response)
Description: Tumors will be assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase by computed tomography (CT) or magnetic resonance imaging (MRI) of target and non-target lesions in accordance with Response Evaluation Criteria in Solid Tumors (irRC) Version 1.1. Percent of subjects with confirmed complete Response or partial response by irRC.
Time Frame: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
Number analyzed (Participants) | 9
Participants | 6

4. Secondary Outcome: Progression Free Survival by RECIST v1.1
Description: PFS were defined as the time from the date of first treatment to the date of disease progression or death (any cause), whichever occured first. Subjects completing study follow-up or starting a new anticancer therapy prior to documented PD were censored in the PFS analysis at the last known date the subject was progression free prior to completing follow-up or initiating new therapy.
Time Frame: Tumors were assessed at screening, and tumor response was assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until disease progression or death (any cause) whichever occurred first. Up to 2.5 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
Number analyzed (Participants) | 9
months | 13.7 [2.2 to NA] — Due to the small number of subjects an upper bound on the confidence interval was not able to be calculated

5. Secondary Outcome: Progression Free Survival by irRC
Description: as for outcome 4
Time Frame: Tumors were assessed at screening, and tumor response was assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until disease progression or death (any cause) whichever occurred first.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
Number analyzed (Participants) | 9
months | 14.3 [2.2 to NA] — Due to the small number of subjects an upper bound on the confidence interval was not able to be calculated

6. Secondary Outcome: Duration of Response by RECIST Version 1.1
Description: DOR were evaluated using Kaplan-Meier methods for those subjects with a confirmed response. DOR were defined as the time from the date of first response (PR or CR) to the date of disease progression or death (any cause) whichever occured first. Responding subjects completing study follow-up or starting a new anticancer therapy prior to documented PD were censored in DOR analysis at the last known date the subject was progression free prior to completing follow-up or initiating new therapy.
Time Frame: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
Number analyzed (Participants) | 5
months | 11.4 [4.9 to NA] — Due to the small number of subjects an upper bound on the confidence interval was not able to be calculated

7. Secondary Outcome: Disease Control Rate by RECIST Version 1.1
Description: Disease control was defined as subjects with a confirmed Complete Response (CR), Partial Response (PR), or Stable Disease (SD) lasting for at least 2 months.
  Complete response (CR; disappearance of all target lesions) or partial response (PR; >=30% decrease in the sum of the longest diameter of target lesions) or stable disease (SD; Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD)
Time Frame: Tumors were assessed at screening, and tumor response will be assessed every 8 weeks during the induction phase, and every 12 weeks during the maintenance phase until disease progression. Up to 2.5 years.
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
Number analyzed (Participants) | 9
Participants
  CR | 2
  PR | 3
  SD greater than or equal to 2 months | 2

8. Secondary Outcome: Duration of Response by irRC
Description: as for outcome 6
Time Frame: as for outcome 5
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
Number analyzed (Participants) | 6
months | 11.4 [4.3 to NA] — Due to the small number of subjects an upper bound on the confidence interval was not able to be calculated

9. Secondary Outcome: Disease Control Rate by irRC
Description: Disease control was defined as subjects with a confirmed Complete Response (irCR), Partial Response (irPR), or Stable Disease (irSD) lasting for at least 2 months.
  Complete response (irCR; disappearance of all index lesions) or partial response (irPR; >=100% decrease in the sum of the longest diameter of index lesions with stable non-index lesions or >=50% decrease in the sum of index lesions with absent/stable /progressed non-index lesions) or stable disease (irSD; Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD)
Time Frame: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
Number analyzed (Participants) | 9
Participants
  irCR | 1
  irPR | 5
  irSD greater than or equal to 2 months | 2

10. Secondary Outcome: Overall Survival
Description: OS were evaluated using Kaplan-Meier methods. OS were defined as the time from the date of first treatment to the date of death (any cause). Subjects who are alive at the end of follow-up were censored in the OS analysis at the last known date alive.
Time Frame: Evaluated from screening to death.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
Number analyzed (Participants) | 9
months | 20.2 [2.4 to 45.2]

11. Secondary Outcome: Quality of Life by Patient Reported Outcomes
Description: Functional Assessment of Cancer Therapy-Breast Cancer (FACT-B) instrument on study
Time Frame: Up to 2.5 years
Population: Due to low enrollment, Quality of Life by Patient Reported Outcomes was not summarized. 0 overall number of participants were analyzed. Data not collected.
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 30 days after last dose, up to 2 years or until resolution or stabilization for nonserious grade 3 or 4 AEs and SAEs, whichever is longer up to 2.5 years
Arm/Group | NANT Triple Negative Breast Cancer (TNBC) Vaccine
All-Cause Mortality (participants affected / at risk) | 7/9
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Triple Negative Breast Cancer (TNBC) Vaccine (N=9)
Disease progression (General disorders) | 1
Injection site reaction (General disorders) | 1
Pyrexia (General disorders) | 1
Mastitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NANT Triple Negative Breast Cancer (TNBC) Vaccine (N=9)
Nausea (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 7
Constipation (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 4
Diarrhoea (Gastrointestinal disorders) | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3
Dry mouth (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Toothache (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Anal inflammation (Gastrointestinal disorders) | 1
Cheilitis (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastrointestinal pain (Gastrointestinal disorders) | 1
Lip erythema (Gastrointestinal disorders) | 1
Lip swelling (Gastrointestinal disorders) | 1
Lip ulceration (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 9
Pyrexia (General disorders) | 9
Injection site reaction (General disorders) | 8
Mucosal inflammation (General disorders) | 8
Chills (General disorders) | 4
Chest discomfort (General disorders) | 4
Axillary pain (General disorders) | 2
Chest pain (General disorders) | 2
Influenza like illness (General disorders) | 2
Injection site erythema (General disorders) | 2
Catheter site erythema (General disorders) | 1
Catheter site pain (General disorders) | 1
Disease progression (General disorders) | 1
Feeling cold (General disorders) | 1
Injection site pruritus (General disorders) | 1
Pain (General disorders) | 1
Swelling (General disorders) | 1
Xerosis (General disorders) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 9
Arthropod sting (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Overdose (Injury, poisoning and procedural complications) | 1
Tracheal deviation (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 6
Paraesthesia (Nervous system disorders) | 4
Dysgeusia (Nervous system disorders) | 2
Neuropathy peripheral (Nervous system disorders) | 2
Presyncope (Nervous system disorders) | 1
Burning sensation (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Horner's syndrome (Nervous system disorders) | 1
Neurological symptom (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Vocal cord paralysis (Nervous system disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 7
Alopecia (Skin and subcutaneous tissue disorders) | 5
Dermatitis contact (Skin and subcutaneous tissue disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1
Papule (Skin and subcutaneous tissue disorders) | 1
Petechiae (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 8
Neutropenia (Blood and lymphatic system disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Lymphopenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Muscle atrophy (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Urinary tract infection (Infections and infestations) | 5
Catheter site cellulitis (Infections and infestations) | 1
Herpes simplex (Infections and infestations) | 1
Implant site infection (Infections and infestations) | 1
Mastitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Skin candida (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Vulval abscess (Infections and infestations) | 1
Weight decreased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Transaminases increased (Investigations) | 1
Weight increased (Investigations) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Pharyngeal swelling (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Anxiety (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Nightmare (Psychiatric disorders) | 2
Irritability (Psychiatric disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Hypotension (Surgical and medical procedures) | 2
Flushing (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Lymphoedema (Vascular disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Ear pain (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Eye disorder (Eye disorders) | 1
Photophobia (Eye disorders) | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Pollakiuria (Renal and urinary disorders) | 1
Hepatobiliary disorders (Renal and urinary disorders) | 1
Cholecystitis (Renal and urinary disorders) | 1
Seasonal allergy (Immune system disorders) | 1
Device occlusion (Product Issues) | 1
RED AND PUFFY LIPS (General disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/85/NCT03387085/Prot_SAP_000.pdf